CLINICAL TRIAL: NCT03385616
Title: A Feasibility Study: A Safety Evaluation of the Gala Airway Treatment System on Patients With Chronic Bronchitis in Canada
Brief Title: Gala Treatment for Chronic Bronchitis in Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gala Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CS004
Record Dates: First submitted 2017-12-18; First posted 2017-12-28 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Chronic Bronchitis; COPD
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Treatment with Gala Airway Treatment System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with GATS (Experimental): Gala Airway Treatment System (GATS)
  Interventions: Device: Gala Airway Treatment System

INTERVENTIONS:
Device: Gala Airway Treatment System — The Gala Airway Treatment system is a device-based, energy delivery system that delivers energy to ablate soft tissue such as the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.
  Other Names: GATS

SUMMARY:
Feasibility trial (FIH) to assess the safety and clinical utility in patients with chronic bronchitis in Canada.

DETAILED DESCRIPTION:
The Gala Airway Treatment system is a device-based, energy delivery system that delivers high frequency short duration energy to the airway epithelium and sub-mucosal tissue layers. The energy is delivered via a proprietary catheter through the bronchoscope.

Two sessions of treatment will be delivered one month apart. The right lung is treated at the first treatment session and the left lung is treated at the second treatment session (approximately one month after the right side is treated). Treatment will be delivered by a respiratory physician (interventional pulmonologist) in a tertiary teaching hospital during a bronchoscopic procedure. The bronchoscopy will be delivered during general anaesthesia. It is anticipated that the bronchoscopic procedure will last less than 60 minutes in total. Treatment will be deemed to have been delivered following the successful treatment during the two bronchoscopies.

A third bronchoscopy will be performed three months following the second treatment session where treatment is not delivered but a cryo-biopsy will be taken from the airway sites that have been treated during the two previous bronchoscopic treatment session to evaluate the effect of the treatment on the airways producing excessive mucous.

Subjects will be required to submit to several tests during the study including two CT scans (lung), respiratory function tests, exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with chronic bronchitis for a minimum of two years, where chronic bronchitis is defined clinically as chronic productive cough for three months in each of two successive years in a patient in whom other causes of productive cough have been excluded.
2. Subject has GOLD Stage II chronic obstructive pulmonary disease (COPD) with a preprocedure post-bronchodilator FEV1 of greater than or equal to 30% and less than or equal to 80% of predicted within three months of enrollment.
3. Subject has an FEV1/FVC ration < 0.7.
4. Subject has been treated with Long Acting Beta Agonists (LABAs) or Long Acting Muscarinic Antagonists (LAMAs) or both for three months or more.
5. Subject has a cigarette smoking history of at least ten packs years.
6. Subject in the opinion of the site investigator is able to adhere to and undergo three bronchoscope procedures inclusive of lung biopsies and Gala treatments, and has provided a signed informed consent.

Exclusion Criteria:

1. Subject has active respiratory infection (e.g., common cold, pneumonia, MAI, tuberculosis) or COPD exacerbation within the last three months.
2. Subject has MMRC score greater than or equal to 3.
3. Subject is taking > 10 mg of prednisolone or prednisone per day.
4. Subject has an implantable cardioverter defibrillator or pacemaker.
5. Subject has a history of cardiac arrhythmia within past two years.
6. Subject has abnormal cardiac rhythm at time of procedure.
7. Subject has history of proven lung cancer in last 5 years.
8. Subject has pulmonary nodule or cavity requiring follow-up or intervention unless proven benign and not actively infected (e.g., aspergilloma).
9. Subject has prior lung surgery, such as lung transplant, LVRS, lung implant/prosthesis, metal stent, valves, coils, bullectomy, segmentectomy, or lobectomy. Pneumothorax without lung resection is acceptable. Pleural procedures without surgery are acceptable.
10. Subject has Alpha-1-Antitrypsin (AAT) deficiency.
11. Subject has documented history of asthma diagnosed with onset <30 years of age, clinically significant bronchiectasis or any other significant second lung disease.
12. Subject actively smoked (including tobacco, marijuana, e-cigarettes, vaping, etc.) within the last 6 months.
13. Subject has known airway colonization with resistant organisms including but not limited to pseudomonas, MRSA, B Cepacia, MTB, M abscessus, mucor or any significant fungus.
14. Subject has the inability to walk over 140 meters.
15. Subject has a serious medical condition, such as: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, hypertension, autoimmune disease or uncontrolled gastric reflux.
16. Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).
17. Subject is pregnant, nursing, or planning to get pregnant during study duration.
18. Subject has received chemotherapy within the past 6 months or is expected to receive chemotherapy during participation in this study.
19. Subject is or has been in another clinical investigational study within 6 weeks of baseline.
20. Subject on anticoagulation for cardiovascular indications and is unable to have anticoagulants (i.e., Aspirin, Plavix, Coumadin) withheld for at least seven days prior to bronchoscopy in the opinion of the Investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of serious adverse events associated with the Gala Airway Treatment System through 6 months. | 6 months
  Incidence of serious adverse events associated with the Gala Airway Treatment System through 6 months.

SECONDARY OUTCOMES:
Clinical Utility - Histology | 3 months following bilateral treatment
  Histopathological evidence of change in mucus producing cells within the airway
Clinical Utility - Pulmonary Function | Through end of study (12-months post-bilateral treatment)
  Pulmonary function testing (PFT) utilizing Forced Expiratory Volume (FEV1)
Quality of Life - CAT | Through end of study (12-months post-bilateral treatment)
  COPD Assessment Test (CAT) questionnaire
Quality of Life - SGRQ | Through end of study (12-months post-bilateral treatment)
  St. George Respiratory Questionnaire (SGRQ)
Acute Exacerbations | From 48 hours post procedure through end of study (12 months post-bilateral treatment)
  Detection of acute exacerbations (measured by clinical examination of a suitably qualified physician)
Non-Acute Exacerbations | From 48 hours post procedure through end of study (12 months post-bilateral treatment)
  Detection of non-acute exacerbations (measured by clinical examination of a suitably qualified physician)
Six Minute Walk Test | 6 months post-bilateral treatment
  Change in 6MWT at 6 months compared to baseline

OTHER OUTCOMES:
CASA-Q | Through end of study (12 months post-bilateral treatment)
  Patient reported outcome respiratory questionnaire: Cough and Sputum Assessment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Director — Gala Therapeutics, Inc.
Locations (3):
- Canada (3):
  - St. Paul's Hospital Vancouver Centre for Heart Lung Innovation, Vancouver, British Columbia
  - Notre Dame Hospital at CHUM, Montreal
  - IUCPQ Quebec, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krimsky WS, Mammarappallil JG, Kim V, Bannan B, Charbonnier JP, Hatton BA, Sciurba FC. Airway Mucus Plugging in Chronic Bronchitis and the Impact of Bronchial Rheoplasty. Chest. 2026 Jan;169(1):73-83. doi: 10.1016/j.chest.2025.06.022. Epub 2025 Jun 24. PMID 40571054